CLINICAL TRIAL: NCT03073122
Title: The Boston Circulatory Arrest Study: Antecedents and Correlates of Well-Being in Adults With Congenital Heart Disease
Acronym: BCAS-Adult
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Gurvitz, Assistant Professor, Boston Children's Hospital
Other Study IDs: P00023574; 1R01HL135061-01 (NIH)
Record Dates: First submitted 2017-01-03; First posted 2017-03-08 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Transposition Great Arteries; Executive Dysfunction
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TGA Case: Brain MRI, Neurocognitive and psychological testing
  Interventions: Diagnostic Test: Brain MRI, neurocognitive and psychological testing
- Control: Brain MRI, Neurocognitive and psychological testing
  Interventions: Diagnostic Test: Brain MRI, neurocognitive and psychological testing

INTERVENTIONS:
Diagnostic Test: Brain MRI, neurocognitive and psychological testing — MRI of the brain and multiple tests of neurocognitive and psychological function including executive function, anxiety and depression

SUMMARY:
In the landmark Boston Circulatory Arrest Study, neurologic and developmental status was measured following infant heart surgery and then prospectively at ages 1, 2.5, 4, 8, and 16 years, with findings of significant neurocognitive deficits and brain MRI abnormalities regardless of operative management. To date, no study has evaluated the neuropsychological and neuroimaging antecedents and correlates of well-being in adults with congenital heart disease, a population now >1 million and projected to grow at 5% per year. The investigators propose to study the Boston cohort at ages 24-29 years to assess the associations of adult well-being with childhood and adolescent executive function, other measures of mental health and cognitive function, adolescent brain MRI findings, and clinical variables; findings will guide the design of interventions in childhood to optimize outcomes in adults with congenital heart disease.

DETAILED DESCRIPTION:
Previously lethal, critical congenital heart disease (CHD) can now be treated effectively with surgical, catheter, and medical interventions. The resulting dramatic improvement in life expectancy has brought a major demographic shift, so that adult patients with CHD now outnumber children with CHD, even for complex conditions. Adult survivors are at increased risk of anxiety, depression, social difficulties, lower educational attainment, and underemployment. These psychosocial morbidities may be associated with deficits in executive functions (EFs) and other neurocognitive abilities that are prevalent in children and adolescents with CHD. Deficits in EFs, represented by measures of inhibitory control, working memory, cognitive flexibility, and decision-making, are highly dependent on the integrity of cortical and subcortical neural networks that continue to develop into early adulthood and can have a major adverse impact on self-regulation and management. The goal of this proposal is to bridge the gap in knowledge between known executive function deficits in childhood CHD and adult well-being. The investigators propose to accomplish our goal by studying subjects, now age 24-29 years, who were enrolled as infants in the Boston Circulatory Arrest Study and then studied with respect to neuropsychological and developmental function at ages 1, 2.5, 4, 8, and 16 years, as well as with brain MRI at 16 years. In Aim 1, the relationship of EFs to major dimensions of adult well-being will be explored. It is hypothesized that lower performance on EFs will be related to poorer overall well-being. The outcomes measured to determine well-being will be quality of life, neuropsychological function (e.g. social cognition, memory skills), mental health diagnosis and function (e.g. anxiety, depression), social relatedness, academic achievement, and adult independence (e.g. employment status, medical follow up). In Aim 2, the relationship of EFs to MRI-derived measures of brain structure, function, and connectivity will be determined. It is hypothesized that lower performance on EFs will be associated with lower global efficiency (integration) and higher modularity (segregation). The brain MRI outcomes will be measured using global white matter connectivity, regional cortical gray matter thickness, gray matter connectivity measured from interregional correlation in cortical thickness, and functional connectivity as defined by resting state functional magnetic resonance imaging. In Aim 3, longitudinal models will be used to analyze the association of adult well-being with earlier measures of EFs and other neurocognitive and mental health variables, as well as with earlier clinical variables and adolescent neuroimaging. The associations of adult well-being dimensions with childhood and adolescent EFs, other measures of mental health and cognitive function, adolescent brain MRI findings, and clinical variables will be explored. The ultimate goal is to identify early, modifiable risk factors for adult performance to guide the design of targeted treatment strategies that optimize educational achievement, employability, and quality of life in the burgeoning population of adults with CHD.

ELIGIBILITY:
Study Group:

Inclusion Criteria

1. Prior participation in the Boston Circulatory Arrest Study
2. Informed consent

Exclusion Criteria

1. Disorders that would prevent successful completion of the planned study testing (severe developmental impairment to prevent answering surveys and participating in interviews)
2. Participants lack of reading fluency in English, which is the only language for which we have the ability to do neuropsychology testing, and for which questionnaires have been validated
3. Women who are currently pregnant will be excluded from the MRI portion of the study only

Control Group:

Control Inclusion Criteria

1. Age 24-30 years at the time of enrollment
2. Informed consent

Control Exclusion Criteria

1. Conditions that would prevent successful completion of the planned study testing (MRI) (e.g., pacemaker, metal implants, orthodontia)
2. Congenital heart disease requiring surgical correction
3. Lack of reading fluency in English, the only language for which questionnaires have been validated
4. Because we purposefully wish to compare d-TGA patients with those in optimal neurodevelopmental health, we will use the exclusion criteria for the NIH-funded project, "MRI study of normal brain development."
5. Current pregnancy

Ages: 24 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Group: All children enrolled in the original boston circulatory arrest study who are alive and living in the US will be invited to participate. We estimate that about 165 adults will be eligible to participate as we will again attempt to contact those patients who did not participate in the 16 year follow-up.
  Controls (for MRI): A group of 50 normally-developed age- and sex-matched young adults ages 24-30 years old who are able to provide informed consent to undergo the MRI portion of the study and limited neuropsychiatric (NP) evaluation. These controls will be recruited from the local metro-Boston area and we will frequency-match control patients to study patients by gender, integer age and handedness.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life health related | baseline
  Linear analog scale, Quality of Life Survey

SECONDARY OUTCOMES:
Mental health - Anxiety | baseline
  Hospital Anxiety and Depression scale and the structured clinical interview for DSM-V
Mental Health - Depression | baseline
  Hospital Anxiety and Depression scale and the structured clinical interview for DSM-V
Mental health - ADHD | baseline
  structured clinical interview for DSM-V and Connors' Adult ADHD Rating Scales - Screening Version
Mental health - PTSD | baseline
  structured clinical interview for DSM-V
Mental health - Stress | baseline
  1. The Stress & Self-Efficacy (Perceived Stress; Self-Efficacy) subdomain of the NIH Toolbox Emotion Domain
Neurocognitive - Executive function | baseline
  1. The Delis-Kaplan Executive Function System (D-KEFS) includes nine subtests: Trail-Making, Verbal Fluency, Design Fluency, Color-Word Interference, Card Sorting, Twenty Questions, Word Context, Tower, and Proverb.
  2. The NIH Toolbox Assessment of Neurological and Behavioral Function, executive function battery is a set of computerized assessments that measure: (a) Inhibitory control (Flanker Inhibitory Control and Attention Test); (b) Working Memory (List Sorting Working Memory Test); (c) Cognitive Flexibility (Dimensional Change Card Sort Test).
  3. The NIH Toolbox Processing Speed assesses the time it takes to process a set amount of information. It yields a main endpoint score.
  4. The Behavior Rating Inventory of Executive Function for Adults (BRIEF-A) includes 75 items that yield 9 clinical scales grouped into two indexes: Behavioral Regulation and Metacognition.
Neurocognitive - Risk taking behavior | baseline
  Iowa Gambling Task (IGT)
Neurocognitive - social cognition | baseline
  1. The "Reading the Mind in the Eyes" Task (revised) is a computer-administered task assessing mental state attribution.
  2. The Advanced Clinical Solutions for WAIS-IV and WMS IV (ACS) is a set of tasks that assess aspects of social cognition, such as affect labeling, affect recognition from faces and prosody, identification of sarcasm, and the ability to verbalize intent of a speaker.
  3. The Autism Spectrum Quotient is a self-report questionnaire covering five domains of autism spectrum disorder: social skills, communication skills, imagination, attention to detail, and attention switching/tolerance of change
Neurocognitive - memory | baseline
  1. The NIH Toolbox Picture Sequence Memory Test evaluates episodic memory.
  2. The Wechsler Memory Scale IV (WMS-IV) provides a comprehensive evaluation of memory abilities in adults, including auditory, visual, immediate, and delayed memory
mental health - social relatedness | baseline
  The NIH Toolbox Emotion Domain - The Social Relationships subdomain measures will be administered.
Employment status | baseline
  Categories from the National health interview survey and Hollingshead four factor index

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gurvitz, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No